CLINICAL TRIAL: NCT00006344
Title: A Randomized, Phase III Dose Response Study of Prophylactic Cranial Irradiation (PCI) for Small Cell Carcinoma of the Lung
Brief Title: Radiation Therapy in Preventing Brain Metastases in Patients With Small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Brian Kavanagh, MD, Virginia Commonwealth University/Massey Cancer Center
Model: Parallel | Purpose: Treatment
Other Study IDs: CDR0000068152; P30CA016059 (NIH); MCV-MCC-9912-2A; NCI-V00-1613
Record Dates: First submitted 2000-10-04; First posted 2004-05-24 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer; extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known which regimen of radiation therapy may be more effective in preventing brain metastases.

PURPOSE: Randomized phase III trial to study the effectiveness of radiation therapy in preventing brain metastases in patients who have small cell lung cancer that has been diagnosed within the past year.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of low dose versus high dose prophylactic cranial irradiation in preventing brain metastases in patients with small cell carcinoma of the lung. II. Determine the neuropsychiatric status of these patients before and after treatment.

OUTLINE: This is a randomized, multicenter study. The right or left hemisphere of each patient's brain are randomized to one of two treatment arms. All patients receive whole brain radiotherapy 5 days a week over 2.5 weeks for a total of 12 fractions. Arm I: Patients receive radiotherapy to the left cerebral hemisphere daily for 6 days immediately following completion of whole brain radiotherapy. Arm II: Patients receive radiotherapy to the right cerebral hemisphere daily for 6 days immediately following completion of whole brain radiotherapy. Patients with extensive disease may also receive thoracic radiotherapy, if not administered previously. Patients are followed at 1, 3, 6, 9, and 12 months, and then every 6 months thereafter.

PROJECTED ACCRUAL: Approximately 16-40 patients will be accrued for this study within 1-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed small cell carcinoma of the lung diagnosed within the past year Limited stage Must have completed prior chemotherapy with thoracic irradiation Extensive stage Must have completed prior chemotherapy with or without thoracic irradiation No more than 24 Gy of prior prophylactic cranial irradiation to the whole brain No brain metastases

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Karnofsky 50-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other prior malignancy within the past 3 years except the following: Adequately treated basal cell or squamous cell skin cancer Carcinoma in situ of the cervix Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-05; Primary Completion 2000-12 (Actual); Study Completion 2000-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kavanagh, MD, Study Chair — Massey Cancer Center
Locations (1):
- Massey Cancer Center, Richmond, Virginia, United States